CLINICAL TRIAL: NCT02877732
Title: EYE-TRAC Advance: Technology Verification (ETA-TV) Cohort 2
Acronym: ETA-TV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The funding sponsor elected to terminate the study.
Sponsor: Stanford University (Other)
Collaborators: Brain Trauma Foundation (Other); United States Department of Defense (U.S. Federal Agency); Food and Drug Administration (FDA) (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jamshid Ghajar, Clinical Professor of Neurosurgery, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20160727
Record Dates: First submitted 2016-08-09; First posted 2016-08-24 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Eye-tracking
Keywords: Concussion; Athletes; Eye-tracking; Vision
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concussed Subject (Experimental): EYE-SYNC eye-tracking device, Level of Alertness, SCAT-3 subtests (Symptom, Immediate memory, Balance and Orientation), Simple Reaction Time subtest of ANAM-SRT and DEM. Investigators will be collecting medical history and demographics from each subject.
  Interventions: Device: EYE-SYNC eye-tracking; Other: SCAT-3 subtests; Other: DEM; Other: Simple Reaction Time subtest of ANAM-SRT; Other: Level of Alertnesss
- Control Subject (Active Comparator): EYE-SYNC eye-tracking device, Level of Alertness, SCAT-3 subtests (Symptom, Immediate memory, Balance and Orientation), Simple Reaction Time subtest of ANAM-SRT and DEM. Investigators will be collecting medical history and demographics from each subject.
  Interventions: Device: EYE-SYNC eye-tracking; Other: SCAT-3 subtests; Other: DEM; Other: Simple Reaction Time subtest of ANAM-SRT; Other: Level of Alertnesss

INTERVENTIONS:
Device: EYE-SYNC eye-tracking — The EYE-SYNC® portable eye-tracking system. The eye tracker is a handheld isolated display environment with embedded eye tracking sensors. The eye tracker is connected to a high-performance Windows tablet though a customized docking station. Included accessories with EYE-SYNC are a U.S. tablet power supply adapter and disposable sanitary masks. Participants are asked to follow a dot with their eyes, as the dot moves on the screen of the EYE-SYNC device.
Other: SCAT-3 subtests — Following subtests of SCAT-3 will be administered to the participant: Symptom, Balance, Orientation and Immediate memory
  Other Names: Sport Concussion Assessment Tool
Other: DEM — Participant will be asked to read list of numbers out loud from a card
  Other Names: Developmental Eye Movement
Other: Simple Reaction Time subtest of ANAM-SRT — Participants will perform Simple Reaction Time sub-test of ANAM-SRT test. They will be asked to click the mouse button every time they see an asterisk on the screen. Participants will perform ANAM-SRT 1 and ANAM-SRT 2 in this study.
  Other Names: Automated Neuropsychological Assessment Metrics
Other: Level of Alertnesss — Participants will answer questions. This assessment is to assess their alertness level.

SUMMARY:
This is a prospective multi-center cohort feasibility and exploratory study.

DETAILED DESCRIPTION:
Investigators propose to prospectively study a cohort of 18-25-year-old athletes to establish the reliability of EYE-SYNC data and the utility of the EYE-SYNC eye-tracking device as a sideline concussion assessment tool. The clinical research study will be conducted to 1) determine if eye-tracking, assessed on the sideline by EYE-SYNC eye-tracking device, is a potential marker of injury that can be used in conjunction with other sideline evaluations to inform decisions regarding removal of athletes from play and 2) to use the EYE-SYNC goggle data as a post- injury recovery monitor.

ELIGIBILITY:
Inclusion Criteria:

Both CCS and CTR must meet the following 3 criteria:

* Athletes between the age of 18- 25-years-old.
* 20/30 or better eyesight (corrected vision allowed).
* English fluency.

Control Subject:

• Control Subject (CTR) - a teammate of the concussed subject who did not experience impact but who was actively participating in the same sport and session along with the injured teammate at the time of injury

Concussed Subject:

Concussed Subject (CCS) - those who experience impact where concussion is highly suspected as evidenced by impairment in any of the SCAT-3 Domains: Symptoms, Physical Signs, Immediate Memory and Orientation. An Injured Athlete is concussed if he/she is FAIL on the Physical Signs, Score = 0 on the Orientation or Scoring below the cutoff scores on the Symptom Checklist and/or Immediate memory SCAT-3 domains.

A) Symptoms: Rating of 2 or higher on any of the following items:

1. Headaches
2. Nausea or Vomiting
3. Dizziness
4. Balance Problems
5. Blurred Vision
6. Feeling Slowed Down
7. Feeling like "in a fog"
8. "Don't feel right"

B) Physical Signs:

Balance (Leg Stances): Number of Error(s) on any of the following 7 subtests classifies a subject as concussed.

I. Double Leg Stance: At least 3 errors II. Single Leg Stance: At least 3 errors with either dominant or non-dominant foot III. Tandem Stance: At least 3 errors or more.

Balance (Tandem Gait): FAIL on at least 2 of 4 trials:

I. FAIL per trial: more than 14 seconds to complete a trial II. FAIL per trial, if one or more of the following errors are made

1. If step off the line;
2. Separation between heel and toe
3. Touch/grab the examiner or an object

D) Orientation: Score = 0 on any of the following 5 items Date: Score = 0 (any date different from current) Month: Score = 0 (any month different from current) Day of the week: Score = 0 (any different from current) Year: Score = 0 (any different from current) Time: Score = 0 AND answer is MORE than + or - 1 hour apart from the correct time.

E) Immediate Memory Recall Total Score = less than 13 words recalled.

Exclusion Criteria:

* Clinical diagnosis of a neurological condition including the following: Stroke, Multiple Sclerosis, Epilepsy, Brain Tumor/Cancer, Nystagmus and/or Other major neurological condition.
* Clinical diagnosis of any of the following eye-sight abnormalities: Uncorrected Amblyopia, Uncorrected Myopia, Uncorrected Presbyopia, Uncorrected Farsightedness, or Uncorrected Astigmatism.
* Psychiatric history with any of the following:

  1. Clinical diagnosis of a psychotic disorder, bipolar disorder - lifetime
  2. Clinical diagnosis of ADHD or ADD - Lifetime
  3. Clinical diagnosis of major depressive disorder - within last year
  4. Clinical diagnosis of substance abuse disorder - within last year
  5. Clinical diagnosis of major anxiety disorder - within last year

     MEDICATION
  6. Requires use of a psychotropic medication.
* Cannot have participated previously in any of the ETA-TV study visits (for instance, a subject that has completed any study visit as a control subject cannot participate as a concussed subject at a later time point).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Little, PhD, Principal Investigator — Stanford University
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - University of California Santa Barbara, Santa Barbara, California
  - Oregon State University, Corvallis, Oregon
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Concussed Subject; Control Subject: EYE-SYNC eye-tracking device, Level of Alertness, SCAT-3 subtests (Symptom, Immediate memory, Balance and Orientation), Simple Reaction Time subtest of ANAM-SRT and DEM.
Period: Overall Study
Arm/Group | Concussed Subject | Control Subject
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concussed Subject | Control Subject | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 20 [18 to 23] | 20 [18 to 23] | 20 [18 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Measurement of EYE-SYNC Data Immediately After Concussive Event, 2 Days, 7 Days and 14 Days Post Concussive Event.
Description: The EYE-SYNC test will be performed immediately after an impact, 2 days, 7 days and 14 days post impact. The movement of eye will be tracked using EYE-SYNC. The data will be recorded in a surface tablet connected to EYE-SYNC.
Time Frame: Immediate post impact, 2 days, 7 days and 14 days post impact.
Population: Study was cancelled by the funder prior to collection of any outcome data; only screening procedures were performed.
Arm/Group | Concussed Subject | Control Subject
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Reliability of EYE-SYNC Data
Description: The integrity will be analyzed based on the score obtained from EYE-SYNC device.
Time Frame: Immediate post impact, 2 days, 7 days and 14 days post impact.
Population: Study was cancelled by the funder prior to collection of any outcome data; only screening procedures were performed.
Arm/Group | Concussed Subject | Control Subject
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Integrity of EYE-SYNC Data
Description: The reliability will be analyzed based on the score obtained from EYE-SYNC.
Time Frame: Immediate post impact, 2 days, 7 days and 14 days post impact.
Population: Study was cancelled by the funder prior to collection of any outcome data; only screening procedures were performed.
Arm/Group | Concussed Subject | Control Subject
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Compare Sport Concussion Assessment Tool (SCAT-3) Test and EYE-SYNC Score
Description: The SCAT-3 result and EYE-SYNC score will be compared.
Time Frame: Immediate post impact, 2 days, 7 days and 14 days post impact.
Population: Study was cancelled by the funder prior to collection of any outcome data; only screening procedures were performed.
Arm/Group | Concussed Subject | Control Subject
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Compare ANAM-SRT Test and EYE-SYNC Score
Description: The Automated Neuropsychological Assessment Metrics-Simple Reaction Time (ANAM-SRT) evaluation and EYE-SYNC score will be compared.
Time Frame: Immediate post impact, 2 days, 7 days and 14 days post impact.
Population: Study was cancelled by the funder prior to collection of any outcome data; only screening procedures were performed.
Arm/Group | Concussed Subject | Control Subject
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Compare DEM Test and EYE-SYNC Score
Description: The Developmental Eye Movement (DEM) assessment and EYE-SYNC score will be compared.
Time Frame: Immediate post impact, 2 days, 7 days and 14 days post impact.
Population: Study was cancelled by the funder prior to collection of any outcome data; only screening procedures were performed.
Arm/Group | Concussed Subject | Control Subject
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study was cancelled by the funder prior to collection of any outcome data; only screening procedures were performed. Adverse Event data was not collected
Description: Study was cancelled by the funder prior to collection of any outcome data; only screening procedures were performed. Adverse Event data was not collected
Arm/Group | Concussed Subject | Control Subject
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT02877732/Prot_SAP_000.pdf